CLINICAL TRIAL: NCT02600312
Title: Comparing Cytokines, Toxins Adsorbing oXiris Filter to ST150 Filter During CRRT in Patients With Septic Shock
Acronym: oXiris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Marcus Broman, M.D. Ph.D., Skane University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: oXiris
Record Dates: First submitted 2015-10-30; First posted 2015-11-09 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oXiris (Active Comparator): Continuous renal replacement therapy with filter that adsorbs cytokines/toxins.
  Interventions: Device: oXiris
- ST150 (No Intervention): Continuous renal replacement therapy with filter that does not adsorb cytokines/toxins.

INTERVENTIONS:
Device: oXiris — oXiris CRRT filter which adsorbs cytokines, toxins.
  Arms: oXiris

SUMMARY:
The Oxiris® filter is a registered product for CRRT already safely used in routine care.

In in vitro experiments, the Oxiris® filter has been demonstrated to adsorb endotoxin and cytokines. Compared to conventional filters this may be advantageous in patients with severe sepsis but neither decreased levels of endotoxin and cytokines nor an improved outcome has been demonstrated with clinical use.

But there are so far little clinical data on the oXiris® filter on humans. The oXiris® filter will be investigated in a double blind randomized crossover setting against a traditional filter (ST150). Either filter will be used for 24 hours after which it will be changed to the opposite filter for another 24 hours.

Arterial blood samples will be drawn at start and then 1, 3, 8, 16 and 24 hours after the start of each filter, and analyzed for endotoxin (EAA assay), TNF-α, IL-1β, IL-6 and IL-10 (ELISA) levels. Standard blood tests will be analyzed simultaneously. Data concerning mode and settings of CRRT, heart rate, blood pressure, medication, data concerning ventilatory support and pathogen will be registered.

Primary endpoint: Levels of endotoxin and cytokines will be compared using Student's paired t-test on AUC values for each 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to intensive care unit (ICU) of age >18 years with decision based on the clinical situation of the patient taken by the physician in charge that continuous renal replacement therapy will be started.
2. Vasoconstrictor and volume dependent septic shock with known Gram-negative infectious agent in blood culture.
3. Vasoconstrictor and volume dependent septic shock suspected to be caused by a Gram-negative agent and with positive plasma endotoxin test.

Exclusion Criteria:

1. Infected with Hepatitis B or C or HIV.
2. Dependence on dialysis treatment before the actual ICU episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
endotoxin level in blood | change from baseline to 48 hours
  Describes the load of toxins from the septic state. Higher load means increased impact from the infectious state mediated through the septic shock.
  Expected mean differences in endotoxin levels including standard deviation is based on data from a previous study on extracorporeal endotoxin removal in sepsis patients (reference 1).

SECONDARY OUTCOMES:
mean blood pressure | hourly up to 48 hours
  Additional parameter that describes the clinical impact from the septic state.
TNF-α level in blood | change from baseline to 48 hours
  Additional parameter that describes the load from the septic shock.
IL-1β level in blood | change from baseline to 48 hours
  Additional parameter that describes the load from the septic shock.
IL-6 level in blood | change from baseline to 48 hours
  Additional parameter that describes the load from the septic shock.
IL-10 | change from baseline to 48 hours
  Additional parameter that describes the load from the septic shock.

OTHER OUTCOMES:
level of vasoconstrictive infusion | hourly up to 48 hours
  Need of vasoconstrictor because of shock, higher degree of shock means increased requirement of vasoconstrictor infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Broman, Associate professor, Principal Investigator — Dep Perioperative and Intensive Care, Skåne University Hospital, Lund, Sweden
Locations (1):
- Perioperative and Intensive Care (Adult), Skåne University Hospital, Lund, Lund, Skåne County, Sweden

REFERENCES:
- [Result] Ala-Kokko TI, Laurila J, Koskenkari J. A new endotoxin adsorber in septic shock: observational case series. Blood Purif. 2011;32(4):303-9. doi: 10.1159/000330323. Epub 2011 Sep 2. PMID 21893976
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356